CLINICAL TRIAL: NCT01384188
Title: A Two-part, Crossover Study to Investigate the Effects of Morning Versus Evening Dosing and Food Interaction on the Pharmacodynamics and Pharmacokinetics of Single and Multiple Doses of ONO-5334 in Healthy Post Menopausal Women
Brief Title: A Study to Investigate the Effects of Food and Morning Versus Evening on Single and Multiple Doses of ONO-5334 in Healthy Post Menopausal Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ONO-5334POE010; 2010-018282-36 (EudraCT Number)
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Post Menopausal Women
MeSH Terms: interventions — ONO-5334

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- E1 (Experimental): ONO-5334
  Interventions: Drug: ONO-5334
- E2 (Experimental): ONO-5334
  Interventions: Drug: ONO-5334

INTERVENTIONS:
Drug: ONO-5334 — 150 mg for 5 days administered in the morning or in the evening
  Arms: E1
Drug: ONO-5334 — 150 mg QD for one day. Administered either in the fasted state or after the standard meal or high fat meal.
  Arms: E2

SUMMARY:
The study will investigate the effects on pharmacodynamics and pharmacokinetics of food and morning versus evening on single and multiple doses of ONO-5334 in healthy post menopausal women.

DETAILED DESCRIPTION:
This study consists of 2 parts. Part 1; The study will investigate the effects of morning versus evening dosing on the pharmacodynamics of multiple doses of 150 mg of ONO-5334 in healthy post menopausal women. The study design will be single-blind and 16 subjects will be enrolled. Part 2; The study will investigate the effects of food on the pharmacokinetics of a single dose of 150mg of ONO-5334 in healthy post menopausal women. 12 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Healthy caucasian women aged between 55 to 75 years inclusive
* Subjects weighing at least 50 kg with mass index between 19 to 30 kg/m2 inclusive
* Subjects who have been amenorrhoeic for at least 5 years.
* Subjects who are confirmed at Screening Visit to have oestradiol and follicle stimulating hormone (FSH) levels consistent with menopause

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of any clinically significant disease or disorder
* Subjects who have a clinically relevant history of insomnia or sleep disorders

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Part 1: Compare pharmacodynamic effect (i.e. urine CTX) of morning versus evening multiple dosing of ONO-5334 | end of treatment (5 days)
Part 2: Compare the effects of food on the pharmacodynamics (i.e., AUC, Cmax) of a single dose of ONO-5334 | end of day 1

SECONDARY OUTCOMES:
Safety and tolerability of single or multiple dose of ONO-5334 in healthy post menopausal women | up to the day after the last dose (Part 1: 5 day multiple doses; Part 2: single dose)

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma UK LTD, Study Director — Ono Pharmaceutical Co. Ltd
Locations (2):
- United Kingdom (2):
  - Guildford Clinical Site, Guildford, Surrey
  - London Clinical Site, London

REFERENCES:
- [Derived] Eastell R, Dijk DJ, Small M, Greenwood A, Sharpe J, Yamada H, Yuba M, Tanimoto M, Deacon S. Morning vs evening dosing of the cathepsin K inhibitor ONO-5334: effects on bone resorption in postmenopausal women in a randomized, phase 1 trial. Osteoporos Int. 2016 Jan;27(1):309-18. doi: 10.1007/s00198-015-3342-4. Epub 2015 Oct 7. PMID 26446770